CLINICAL TRIAL: NCT04944693
Title: A Prospective Study of Anterior Tibial Subluxation in the Setting of Anterior Cruciate Ligament Reconstruction With 2-year Follow-up
Brief Title: Relationship Between Anterior Tibial Subluxation and the Prognosis of Anterior Cruciate Ligament Reconstruction.
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020384
Record Dates: First submitted 2021-06-27; First posted 2021-06-29 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior tibial subluxation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Anterior cruciate ligament-injured patients with excessive ATS
  Interventions: Other: Different ATS values.
- Cohort 2: Anterior cruciate ligament-injured patients with minimal ATS
  Interventions: Other: Different ATS values.

INTERVENTIONS:
Other: Different ATS values. — Observational, different ATS values were measured on MRI images and were regarded as "interventions" for different cohorts.

SUMMARY:
To identify the improvement of anterior tibial subluxation (ATS) and the relationship between ATS and patient reported outcome on pre- and postoperative anterior cruciate ligament-injured MRI images.

DETAILED DESCRIPTION:
The value of preoperative anterior tibial subluxation (ATS) was used for the division of anterior cruciate ligament-injured patients in 2 groups. ATS was measured on pre- and postoperative MRI images. Patients were followed up 2 years after anterior cruciate ligament reconstruction, and patient reported outcomes (i.e. Lysholm score, etc.) were collected for further analysis.

ELIGIBILITY:
Inclusion Criteria: (1) Diagnosed anterior cruciate ligament injuries; (2) available preoperative MRI scans at our hospital.

-

Exclusion Criteria: Patients were excluded in the case of under 18 years of age, bilateral anterior cruciate ligament injuries, concomitant posterior cruciate ligament injuries, concomitant collateral ligament injuries, and no access to the preoperative MRI scan at our hospital.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: anterior cruciate ligament-injured patients that had suffered from anterior cruciate ligament injury.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Patients reported outcomes | at least 1-year postoperatively
  (i.e. Lysholm score, etc.)

SECONDARY OUTCOMES:
MRI images | at least 1-year postoperatively
  Anterior tibial subluxation were measured on postoperative MRI images

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No